CLINICAL TRIAL: NCT01697735
Title: The Therapeutic Effects of Combination of Statins With Berberine on the Patients With Hyperlipemia:a Single-center, Open Clinical Trial
Brief Title: The Therapeutic Effects of Statins and Berberine on the Hyperlipemia
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Because of lack of participants and funds
Sponsor: Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, Kangting Ji, MD, Director, Wenzhou Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: WZ medical college
Record Dates: First submitted 2012-09-28; First posted 2012-10-02 (Estimated); Last update posted 2016-04-28 (Estimated); Status verified 2016-04

CONDITIONS: Dyslipidemias
MeSH Terms: conditions — Dyslipidemias | interventions — Rosuvastatin Calcium; Berberine; Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Berberine;Atorvastatin or Rosuvastatin (Experimental): Follow the previous administration program，participants will continue to receive 20mg Atorvastatin daily or 10mg Rosuvastatin daily; Besides taking statins, Participants will receive 500mg berberine twice a day for 8 weeks.
  Interventions: Drug: Berberine;Atorvastatin or Rosuvastatin
- Atorvastatin or Rosuvastatin (Active Comparator): Due to the different clinical prescriptions by different doctors and similar Efficacy in lowering lipids.Usually,Participants receive 20mg Atorvastatin daily or 10mg Rosuvastatin to treat hyperlipidemia.
  Interventions: Drug: Atorvastatin or Rosuvastatin

INTERVENTIONS:
Drug: Berberine;Atorvastatin or Rosuvastatin — Participants will receive 500mg Berberine twice a day for 8 weeks; Follow the previous administration program，participants will continue to receive 20mg Atorvastatin daily or 10mg Rosuvastatin daily.
  Other Names: Berberine;; Liptor; Crestor
  Arms: Berberine;Atorvastatin or Rosuvastatin
Drug: Atorvastatin or Rosuvastatin — Due to the different clinical prescriptions by different doctors and similar Efficacy in lowering lipids.Usually,Participants receive 20mg Atorvastatin daily or 10mg Rosuvastatin to treat hyperlipidemia.
  Other Names: Liptor; Crestor
  Arms: Atorvastatin or Rosuvastatin

SUMMARY:
Statins are cholesterol-lowering medications that are often prescribed for patients with high cholesterol and who are at risk for cardiovascular disease (CVD). But there are many patients whose hyperlipemia are not well controlled. If investigators are simply doubling the statins, that only 6% of the benefit can be received. And it often has significant side effects in elder patients. Several studies have suggested that the use of berberine can effectively lower blood lipids. The chemical structure and mechanisms of drug is clearly, and the side effects are seldom, the price of berberine is very cheap. The purpose of this study is to observe the therapeutic effects of combination of statins and berberine on the patients with hyperlipemia whose level of the lipid are not well controlled when only using statins.

DETAILED DESCRIPTION:
Patients at risk for cardiovascular disease (CVD) are often prescribed statins, which are medications that reduce the amount of cholesterol in the blood. By lowering cholesterol levels, these patients have a lower incidence of coronary artery disease, ischemic stroke, and peripheral arterial disease and so on. But there are many patients whose hyperlipemia are not well controlled.If investigators are simply doubling the statins, that only 6% of the benefit can be received.And it often bring significant side effects in elder patients. Several studies have suggested that the use of berberine can effectively lowering blood lipids.The chemical structure and mechanisms of drug is clearly, and the side effects are seldom, the price of berberine is very cheap. The purpose of this study is to observe the therapeutic effects of combination of statins and berberine on the patients with hyperlipemia whose level of the lipid are not well controlled when only using statins.

This study will enroll patients who currently take cholesterol-lowering medications，but the level of lipid is not controlled well. Patients will be assigned to receive 500mg of Berberine twice a day(meanwhile they are taking 20mg of Atorvastatin daily for 8 weeks or 10mg of Rosuvastatin daily for 8 weeks). Investigators will occur at baseline and Weeks 4 and 8. Blood will be collected for laboratory testing, and standardized psychological questionnaires will assess fatigue at baseline and weeks 4 and 8. Pill count will be used to assess adherence of Berberine and statins treatment at weeks 4 and 8. At weeks 4 and 8, medication side effects will be monitored and tests of alanine aminotransferase (ALT) and creatine phosphate kinase (CPK) will be performed. At weeks 4 and 8, medication efficacy will be assessed and test of low-density lipoprotein cholesterol (LDL-C) will be performed.

ELIGIBILITY:
Inclusion Criteria:

1. Current use of lipid-lowering medications;
2. Documented cardiovascular disease (CVD) by invasive or non-invasive testing (such as coronary angiography, nuclear imaging, stress echocardiography, carotid plaque on ultrasound), previous myocardial infarction (MI), acute coronary syndrome (ACS), coronary revascularization [percutaneous coronary intervention (PCI), coronary artery bypass graft (CABG)] and other arterial revascularization procedures, ischaemic stroke, peripheral arterial disease(PAD);
3. Patients with type 2 diabetes, patients with type 1 diabetes with target organ damage (such as microalbuminuria); Patients with moderate to severe chronic kidney disease [glomerular filtration rate (GFR) < 60 mL/min/1.73㎡];
4. Markedly elevated single risk factors such as familial dyslipidaemias and severe hypertension;
5. A calculated SCORE ≥1% for 10 year risk of fatal CVD

Exclusion Criteria:

1. Cancer;
2. HIV infected;
3. Medical or psychiatric condition that prevents full study participation or follow-up (e.g., active psychosis);
4. Active liver disease or unexplained persistent elevated transaminase levels；
5. Major surgery or hospitalization in the 3 months prior to study entry;
6. Current use of cyclosporin, erythromycin, clarithromycin, nefazodone, or any "azole" antifungals, including fluconazole, itraconazole, ketoconazole, mibefradil, or protease inhibitors;
7. Female of childbearing potential;
8. Severe gastrointestinal disease;
9. With berberine using contraindications;
10. Secondary hyperlipidemia
11. Current participation in another clinical trial

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-09; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline in combination statins with berberine on lipid level | Measured at baseline, weeks 4 and 8

SECONDARY OUTCOMES:
Adherence of statins and berberine treatment | Measured at weeks 4 and 8

CONTACTS AND LOCATIONS:
Overall Officials: Jifei Tang, MD, Principal Investigator — Wenzhou Medical University
Locations (1):
- Second Hospital of Wenzhou Medical College, Wenzhou, Zhejiang, China